CLINICAL TRIAL: NCT06839040
Title: Effects of a Multidisciplinary Intervention on Fall Risk and Urinary Incontinence in Older Women
Acronym: FIRE-WOMEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Jorge Alarcón Jiménez, Professor, Fundación Universidad Católica de Valencia San Vicente Mártir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2022-2023/123
Record Dates: First submitted 2025-02-04; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Urinary Incontinence; Frailty; Balance Impairment
Keywords: older women; pelvic floor; balance; multicomponent exercise; urinary incontinence; phsychoeducation
MeSH Terms: conditions — Urinary Incontinence; Frailty

STUDY DESIGN:
Intervention Model Description: This will be a double blind (investigator-evaluator/data analyst), four arm experimental, parallel and longitudinal study.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Multi-component exercise group with verbal instructions for the pelvic floor and psychoeducation (Experimental): A multidisciplinary intervention will be carried out, consisting of an initial phase of individual physiotherapy based on specific active muscle training of the pelvic floor (EMSP). This will be followed by a group-based multi-component physical exercise program with instructions on pelvic floor contraction during the exercises, and psychoeducation sessions to help cope with the fear of increased likelihood of falls and urinary incontinence as a result of aging.
  Interventions: Other: Group 1: ExVerbPsy
- Multi-component exercise group with verbal instructions for the pelvic floor (Active Comparator): The same procedure as experimental group 1 (exercise + verbal instructions + psychoeducation) will be performed except for the psychoeducation sessions.
  Interventions: Other: Group 2: ExVerb
- Multicomponent exercise group without verbal instructions for the pelvic floor (Active Comparator): The same procedure as experimental group 1 (exercise + verbal instructions + psychoeducation) will be performed but without verbal instructions and psychoeducation sessions.
  Interventions: Other: Group 3: Ex
- Control group (No Intervention): They will receive information sessions on the prevention of geriatric syndromes and will be asked to maintain their normal activity level. At the end of the interventions, this group will have the option of receiving the appropriate intervention that was not carried out in the initial process.

INTERVENTIONS:
Other: Group 1: ExVerbPsy — A multidisciplinary intervention will be carried out, consisting of an initial phase of individual physiotherapy based on specific active muscle training of the pelvic floor (EMSP). This will be followed by a group-based multi-component physical exercise program with instructions on pelvic floor contraction during the exercises, and psychoeducation sessions to help cope with the fear of increased likelihood of falls and urinary incontinence as a result of aging.
  Arms: Multi-component exercise group with verbal instructions for the pelvic floor and psychoeducation
Other: Group 2: ExVerb — The same procedure as experimental group 1 ExVerbPsy will be performed except for the psychoeducation sessions.
  Arms: Multi-component exercise group with verbal instructions for the pelvic floor
Other: Group 3: Ex — The same procedure as experimental group 1 ExVerbPsy will be performed but without verbal instructions and psychoeducation sessions.
  Arms: Multicomponent exercise group without verbal instructions for the pelvic floor

SUMMARY:
This will be a quantitative, quasi-experimental, and longitudinal study spanning 18 weeks of intervention, followed by a 24-week follow-up, scheduled to begin in January 2025.

The primary objective of this study is to evaluate the effects of a multidisciplinary intervention comprising physiotherapy, physical exercise, and psychoeducation on fall risk and urinary incontinence in non-institutionalized older adult women aged 60 to 80 years. Participants will be randomly assigned to one of four groups:

1. A multicomponent exercise group with verbal instructions for pelvic floor exercises.
2. A multicomponent exercise group with verbal instructions for pelvic floor exercises and psychoeducation.
3. A multicomponent exercise group without verbal instructions for pelvic floor exercises.
4. A control group.

Multicomponent exercise sessions will be conducted twice a week, while the psychoeducation group will participate in five group therapy sessions throughout the program. The variables to be analyzed include balance, strength, power, pelvic floor function, quality of life, and self-esteem.

DETAILED DESCRIPTION:
The aging process can lead to the development of major geriatric syndromes, such as falls and urinary incontinence. Although there are studies demonstrating the effectiveness of physical exercise and education in addressing these conditions, there is currently very limited evidence on the combined effects of both therapies on these syndromes.

The primary objective of this study is to evaluate the effects of a multidisciplinary intervention consisting of physiotherapy, physical exercise, and psychoeducation on the risk of falls and urinary incontinence in older adult women.

Methods: This will be a quantitative, quasi-experimental, and longitudinal study with 18 weeks of intervention and a 24-week follow-up period. The study is scheduled to begin in January 2025. The sample will consist of non-institutionalized older adult women aged between 60 and 80 years, who will be randomly assigned to one of four groups:

1. A multicomponent exercise group with verbal instructions targeting the pelvic floor.
2. A multicomponent exercise group with verbal instructions targeting the pelvic floor and psychoeducation.
3. A multicomponent exercise group without verbal instructions targeting the pelvic floor.
4. A control group.

Multicomponent exercise sessions will be conducted twice a week and will include exercises focused on balance, strength/power using elastic bands, aerobic capacity, and coordination. The verbal instructions for the pelvic floor will involve performing fast and slow contractions during the general exercises. Participants in the psychoeducation group will attend five group therapy sessions throughout the program.

The study will analyze variables related to balance (Timed Up and Go test, functional reach test, and posturography), lower limb strength/power (isometric strength tests and jump performance), and pelvic floor function (using the PERFECT scale and electromyography). Additionally, physical, psychological, and social well-being variables will be assessed using instruments such as the SF-36, ICIQ-SF, and Rosenberg self-esteem scale.

Results/Conclusion: It is anticipated that differences will emerge between the study groups, with the trimodal intervention group (multicomponent exercise + specific verbal instructions for the pelvic floor + psychoeducation) showing greater improvements in certain parameters.

ELIGIBILITY:
Inclusion Criteria:

* Woman, aged between 60 and 80 years.
* Not having done physical exercise in the last 3 months.
* Present UI (SUI, UUI or MUI) after clinical diagnosis.
* Score greater than 90 on the Barthel Scale.
* Not present pathologies or functional alterations that limit the practice of physical exercise.
* Not present severe cognitive alterations or mild cognitive deficit (Global Deterioration Scale less than or equal to 2 or Mini Mental State Examination greater than or equal to 25 points).
* Maintain walking without support products.
* Carry out 80% of the total sessions

Exclusion Criteria:

* Intake of medication that could affect the performance of the exercise or alter the variables studied.
* Present grade II-IV uterine prolapses.
* Clinical disease or syndrome (chronic or acute cardiovascular, neurological, respiratory or musculoskeletal disorders) that may interfere with the performance of the intervention and evaluation.
* Present visual and/or auditory alterations that make it difficult to carry out the intervention and evaluation.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-02 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor | From enrollment to the end of treatment at 18 weeks
  PERFECT Scale:
  Power (P): with Oxford scale 0 to 5 points Endurence (E): 0 to 10 points Repetitions (R): 0 to 10 points Fast (F): 0 to 10 points
Pelvic floor | From enrollment to the end of treatment at 18 weeks.
  Intracavitary electromyography: maximum and average contraction. Outcome measure in microvolts.
Pelvic floor | From enrollment to the end of treatment at 18 weeks.
  Manometric perineometer: maximum contraction. Outcome measure in millimeters of mercury.
Abdominal muscle tone | From enrollment to the end of treatment at 18 weeks.
  Abdominal ultrasound of rectus and transverse abdominis: in relaxation and activation with diaphragmatic breathing. Outcome measure in milimeters.
Dynamic balance | From enrollment to the end of treatment at 18 weeks
  Timed Up and Go: the time it takes for the person to get up from a chair, walk 3 meters, turn on a cone, return to the chair and sit down. Outcome measure in seconds. Less than 10 seconds: low risk of falling. Between 10 and 20 seconds: frailty (medium risk of falling). More than 20 seconds: high risk of falling and disability.
Static balance | From enrollment to the end of treatment at 18 weeks.
  Romberg test with feet together, semi-tandem and tandem in 10 seconds. Static one-leg standing balance test with open and closed eyes in 30 seconds. Outcome measure in seconds.
Static balance | From enrollment to the end of treatment at 18 weeks.
  Posturography with and without balance foam: anteroposterior and lateral axis oscillation, and degree of shift of the center of gravity (COP). Outcome measure in milimeters.
Static balance | From enrollment to the end of treatment at 18 weeks.
  Functional reach: distance traveled in anterior displacement with arms outstretched and feet together. Outcome measure in centimeters.
Gait | From enrollment to the end of treatment at 18 weeks
  Six minutes gait with Runscribe sensors on feet and four meters gait (normal and fast speed)
Power | From enrollment to the end of treatment at 18 weeks
  Jumps (CMJ and ABK), leg extension and squad. Outcome measure in wats.
Power and strenght | From enrollment to the end of treatment at 18 weeks
  Five sit to stand, thirty sit to stand and arm curl. Outcome measure in number of repetitions in 30 seconds.
Strenght and endurance | From enrollment to the end of treatment at 18 weeks
  Isometries of leg extension, hip extension, hip abduction, hip adduction, spine extension and hand grip. Outcome measure in newtons.
Health impact and quality of life | From enrollment to the end of treatment at 18 weeks.
  International Consultation on Incontinence Questionnaire (ICIQ-SF): 0 to 21 points from urinary incontinence impact. Outcome measure in units on a scale.
Psychological and social well-being | From enrollment to the end of treatment at 18 weeks.
  Falls efficacy scale: 16 to 64 points from least to most worry about falling. Outcome measure in units on a scale.

SECONDARY OUTCOMES:
Quality of live | From enrollment to the end of treatment at 18 weeks
  Quality of live with questionnaire Short Form (SF36): this questionnaire evalues in 36 questions the physical function, physical role, body pain, general health, vitality, social function, emotional role, and mental health. 0 to 100 points. Outcome measure in units on a scale.
Psychological and social well-being | From enrollment to the end of treatment at 18 weeks.
  Self-esteem questionnaire of Rosenberg: 10 points low self-esteem to 40 points high self-esteem. Outcome measure in units on a scale.
Weight | From enrollment to the end of treatment at 18 weeks
  Kilograms and information on percentage of lean mass and fat mass.
Height | From enrollment to the end of treatment at 18 weeks
  Stadiometer. Outcome measure in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: ESTHER RAMOS CASTELLANO, Principal Investigator — Escuela de Doctorado. Universidad Católica de Valencia San Vicente Mártir (Doctoral School. Catholic University of Valencia San Vicente Mártir)
Locations (1):
- Escuela de Doctorado. Universidad Católica de Valencia San Vicente Mártir. (Doctoral School. Catholic University of ValenciaSan Vicente Mártir), Valencia, Valencia, Spain